CLINICAL TRIAL: NCT05205603
Title: Efficacy of Mesalazine Combined With Biologics in the Treatment of Moderate to Severe Ulcerative Colitis: a Multicenter, Prospective, Randomized, Controlled Clinical Study
Brief Title: Efficacy of Mesalazine Combined With Biologics in the Treatment of Moderate to Severe Ulcerative Colitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021ZSLYEC-456
Record Dates: First submitted 2022-01-05; First posted 2022-01-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Ulcerative Colitis; Efficacy, Self; Biologics; Mesalazine
Keywords: ulcerative colitis; biologics; mesalazine
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; vedolizumab; Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biologics group (Placebo Comparator): Biologics including infliximab and vedolizumab. infliximab: 5mg/kg, intravenously administration at week 0, 2, and 6 as induction therapy; subsequently by maintenance therapy at a dose of 5mg/kg every 8 weeks.
  vedolizumab: 300mg, intravenously administration at week 0, 2, and 6 as induction therapy; subsequently by maintenance therapy at a dose of 300mg every 8 weeks.
  Interventions: Drug: Infliximab; Drug: Vedolizumab
- 5-ASA group (Experimental): 5-ASA combined with biologics (including infliximab and vedolizumab). infliximab: 5mg/kg, intravenously administration at week 0, 2, and 6 as induction therapy; subsequently by maintenance therapy at a dose of 5mg/kg every 8 weeks.
  vedolizumab: 300mg, intravenously administration at week 0, 2, and 6 as induction therapy; subsequently by maintenance therapy at a dose of 300mg every 8 weeks.
  mesalazine: at a dose of 4-6g/d systemic or topical therapy
  Interventions: Drug: Infliximab; Drug: Vedolizumab; Drug: Mesalazine

INTERVENTIONS:
Drug: Infliximab — Infliximab, 5mg/kg at week 0,2,6 and schedule administration at every 8 weeks
Drug: Vedolizumab — Vedolizumab, 300mg at week 0,2,6 and schedule administration at every 8 weeks
Drug: Mesalazine — Mesalazine, 4-6g/d, systemic and/or topical administration
  Arms: 5-ASA group

SUMMARY:
Endocopic remission rates of moderate to severe ulcerative colitis are low. Biologics including Vedolizumab, infliximab, and adalimumab are effective in induction and maintainence of ulcerative colitis. The role of 5-ASA in promoting a higher rate of endocsopic remission is unclear. We aim to evaluate the efficacy of combination of 5-ASA and biologics in treating ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate and severe ulcerative colitis;
2. Subjects were above 18 years old and below 80 years;
3. Indications of 5-ASA or biological treatment;
4. According to the clinical symptoms, ulcerative colitis was diagnosed by endoscopic changes, pathological manifestations. The disease activity of UC was assessed according to the modified Mayo scoring system (modified Mayo: 6~12 for patients with moderate to severe ulcerative colitis);
5. If the subject is a woman, a pregnancy test at baseline is needed to exclude pregnancy. Female patients must follow the contraceptive recommendations of the project;
6. Subjects must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

Exclusion Criteria:

1. No indications of 5-ASA or biological treatment;
2. ulcerative colitis patients who had previously undergone a partial colectomy;
3. Patients who are unable to use 5-ASA for a long time;
4. Patients with severe, progressive, or uncontrolled kidney, liver, blood, or endocrine diseases or symptoms;
5. Presence of infected persons, Patients with a contraindication to the use of biological agents such as C. difficile infection or other intestinal pathogens, active tuberculosis or intestinal tuberculosis infection, human immunodeficiency virus (HIV) infection, active hepatitis B or hepatitis C (defined as: ① HBV: hepatitis B surface antigen (HBs Ag) positive (+), Or patients with positive for hepatitis B core antibody (HBcAb) and the qualitative test results of HBV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) meet the detection criteria; ② HCV: Any patient with an anti-HCV antibody (HCV Ab) -positive patient with a detectable HCV ribonucleic acid (RNA);
6. Patients with a history of gastrointestinal dysplasia, or dysplasia on any biopsy performed on endoscopy, excluding low-grade dysplasia lesions; known history of lymphoproliferative disease (including lymphoma), or signs and symptoms (e. g., lymphadenopathy and / or splenomegaly); patients with current or previous malignancy;
7. Has been involved in other clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
endoscopic remission rate at 12 months | 12 months after first intervention administration
  endoscopic remission rate at 12 months

SECONDARY OUTCOMES:
normalization rate of serum biomarker at 12 months | 12 months after first intervention administration
  normalization rate of serum biomarker at 12 months
normalization rate of serum biomarker at 6 months | 6 months after first intervention administration
  normalization rate of serum biomarker at 6 months
clinical remission rate at 12 months | 12 months after first intervention administration
  clinical remission rate at 12 months
clinical remission rate at 6 months | 6 months after first intervention administration
  clinical remission rate at 6 months
clinical response rate at 12 months | 12 months after first intervention administration
  clinical response rate at 12 months
clinical response rate at 6 months | 6 months after first intervention administration
  clinical response rate at 6 months
endoscopic remission rate at 6 months | 6 months after first intervention administration
  endoscopic remission rate at 6 months
endoscopic response rate at 12 months | 12 months after first intervention administration
  endoscopic response rate at 12 months
endoscopic response rate at 6 months | 6 months after first intervention administration
  endoscopic response rate at 6 months
life quality changes at 12 months | 12 months after first intervention administration
  life quality evaluated by IBDQ (inflammatory bowel disease questionnaire) at 12 months
life quality changes at 6 months | 6 months after first intervention administration
  life quality evaluated by IBDQ (inflammatory bowel disease questionnaire) at 6 months

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - First People's Hospital of Foshan, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Nanhai Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shunde Hospital of Southern Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital, Shenyang, Liaoning
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Zhejiang University, Hanzhou, Zhejiang